CLINICAL TRIAL: NCT03397212
Title: Assessment of NADA Acupuncture for Treatment of Withdrawal Symptoms During Gradual Opioid Withdrawal in Chronic Pain Patients
Brief Title: Treatment of Withdrawal Symptoms With NADA Acupuncture in Chronic Pain Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Romanas Polianskis, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 59065
Record Dates: First submitted 2017-11-29; First posted 2018-01-11 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Chronic Pain; Opiate Withdrawal Syndrome
Keywords: NADA
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NADA and Clonidine (Experimental): NADA acupuncture and treatment with tbl Clonidine
  Interventions: Other: NADA acupuncture
- Sham acupuncture and Clonidine (Sham Comparator): Sham ear acupuncture and treatment with tbl Clonidine
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: NADA acupuncture — Ear acupuncture protocol described by National Acupuncture Detoxification Association
  Arms: NADA and Clonidine
Other: Sham acupuncture — Ear acupuncture using inactive sham points
  Arms: Sham acupuncture and Clonidine

SUMMARY:
This project aims at examining the following hypotheses:

* Treatment with NADA and clonidine reduces intensity of withdrawal symptoms to a greater extent than treatment with clonidine.
* Opioid withdrawal improves pain, physical and mental functioning and reduces opioid consumption 3 months and 1 year after withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain patients treated with opioids over 3 months
* The patient's doctor or nurse assesses that there is an indication to opioid withdrawal and / or the patient wishes to withdraw.
* The patient is motivated for opioid withdrawal
* The patient has experienced withdrawal symptoms
* The patient must be able to understand, speak and write Danish
* The patient must be able to transport himself to the pain center

Exclusion Criteria:

* Children under 18 years old
* External ear infection
* Treatment with benzodiazepines.
* Active substance abuse and alcohol abuse.
* Contraindications for treatment with clonidine:
* Allergy
* Bradyarrhythmias caused by diseased sinus cube or AV block of 2nd or 3rd grade.
* lactose intolerance
* Heart failure
* High medullary damage
* Cardiac conduction disturbances
* Pregnancy and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-15 (Estimated); Primary Completion 2022-01-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in intensity of withdrawal symptoms | 3 months and 1 year
  Change in intensity of withdrawal symptoms assessed with Danish withdrawal symptom questionnaire

SECONDARY OUTCOMES:
Change in quality of life assessed with SF36 | 3 months and 1 year
  Change in quality of life assessed with SF36

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No